CLINICAL TRIAL: NCT05248724
Title: Periarticular Injection and Hamstring Block Versus Placebo for Pain Control in Anterior Cruciate Ligament Reconstruction: A Randomized Controlled Trial
Brief Title: Periarticular Injection and Hamstring Block Versus Placebo for Pain Control in Anterior Cruciate Ligament Reconstruction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Castilla-La Mancha Health Service (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2017/PI0217
Record Dates: First submitted 2022-02-06; First posted 2022-02-21 (Actual); Last update posted 2022-03-08 (Actual); Status verified 2022-02

CONDITIONS: Anterior Cruciate Ligament Reconstruction
Keywords: postoperative analgesia; Local Anesthetic; postoperative pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Ropivacaine; Ketorolac Tromethamine; Epinephrine

STUDY DESIGN:
Intervention Model Description: This study was a prospective single-blind, two arms, parallel-group
Who Masked: Participant
Masking Description: The participants were not informed about what group (intervention or placebo) they were assigned.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention, (Experimental): Patients allocated to the intervention group received a periarticular infiltration with a solution containing 200 mg of ropivacaine hydrochloride (10mg/ml Kabi Fresenius Kabi Norway AS),150 mg if the patient weight was below 65kg, 5 mg of morphine hydrochloride (10mg/ml Braun Medical SA Spain), 30 mg of ketorolac tromethamine (Normon Spain), 300 micrograms of adrenaline (epinephrine Braun Medical SA Spain), and saline 0.9% till reaching 50 ml of volume
  Interventions: Combination Product: periarticular infiltration (50ml) with Ropivacaine Hydrochloride 10 MG/ML (200 mg) + ketorolac tromethamine 30 mg/ml (30 mg) + adrenaline 1mg/ml (300 microgram) + morphine hydrochloride 10mg/ml (5 mg)
- placebo (Placebo Comparator): Participants in the placebo group received a periarticular infiltration of 50 ml of saline 0.9%.
  Interventions: Drug: placebo

INTERVENTIONS:
Combination Product: periarticular infiltration (50ml) with Ropivacaine Hydrochloride 10 MG/ML (200 mg) + ketorolac tromethamine 30 mg/ml (30 mg) + adrenaline 1mg/ml (300 microgram) + morphine hydrochloride 10mg/ml (5 mg) — Patients allocated to the intervention group received a periarticular infiltration with a solution containing 200 mg of ropivacaine hydrochloride ,150 mg if the patient weight was below 65kg, 5 mg of morphine hydrochloride , 30 mg of ketorolac tromethamine, 300 micrograms of adrenaline and saline 0.9% till reaching 50 ml of volume. Half of the solution was injected into the proximal hamstring stump. The surgical team closed the wounds and injected the other half of the intervention into the subcutaneous tissue in the distal wound and portals. There was not any medication introduced inside the articulation. Patients of the placebo group were treated in the same way, but the solution injected was 50 ml of saline 0.9%.
  Arms: Intervention,
Drug: placebo — 50 ml of 0.9 saline
  Arms: placebo

SUMMARY:
A randomized controlled trial about periarticular injection and hamstring block versus placebo for pain control in anterior cruciate ligament reconstruction

DETAILED DESCRIPTION:
This study was a prospective, two arms, parallel-group, randomized controlled trial conducted in a single second-level hospital in Spain. The ethics committee of the institution approved the study. Every patient received complete information and signed written consent. A total of 44 patients were randomized in two groups assigned to receive PI or placebo. The perioperative protocol was the same for both groups. The principal outcome was pain measured at 8 and 24 hours by a visual analog scale (VAS). The pain was registered in the knee and the proximal donor site. Pain scores were also assessed to determine whether the VAS improvement would reach the threshold values reported for the minimal clinically significant difference. The secondary outcome was the need for opioid rescue medication.

The surgical procedure was a single bundle transtibial mono tunnel technique with autologous hamstring under limb ischemia.

Patients allocated to the intervention group received a periarticular infiltration with a solution containing 200 mg of ropivacaine hydrochloride (10mg/ml Kabi Fresenius Kabi Norway AS),150 mg if the patient weight was below 65kg, 5 mg of morphine hydrochloride (10mg/ml Braun Medical SA Spain), 30 mg of ketorolac tromethamine (Normon Spain), 300 micrograms of adrenaline (epinephrine Braun Medical SA Spain), and saline 0.9% till reaching 50 ml of volume. The surgical operation nurse prepared the mixture under sterile conditions at the end of the procedure. The 50 ml syringe was connected to a female probe. The surgeon introduced the female probe inside the closed tendon stripper to use it as a guide. The tendon stripper and female probe were inserted through the distal wound to the proximal stump of the hamstring muscles. Half of the solution was injected into this area. The assistant extended the knee, and the sartorius fascia was sutured to minimize the leaking of the mixture. The surgical team closed the wounds and injected the other half of the intervention into the subcutaneous tissue in the distal wound and portals. There was not any medication introduced inside the articulation. Patients of the placebo group were treated in the same way, but the solution injected was 50 ml of saline 0.9%.

The primary outcome was pain registered in the knee and the posterior proximal thigh at 8 and 24 hours from the surgery. The pain was rated using a 100 mm horizontal line, for which 0 represented no pain and 100 maximum pain. In addition to statistical significance, differences in patient-reported outcomes should be assessed for clinical importance or relevance. The secondary outcome was the need for analgesic rescue medication in the post-anesthesia care unit and during the stay in the orthopedics ward. Complications throughout the hospitalization and in the first month were also registered.

All statistical analyses were performed using IBM SPSS 25.0 Statistics software, and the level of significance was set at α < 0.05. Data are presented as mean (standard deviation-SD) for continuous variables and as counts and percentages for categorical variables. Characteristics of participants were compared IP group vs. control group using the Chi-square test for categorical variables and Student's t-test for continuous variables.

ELIGIBILITY:
Inclusion Criteria:

* Anterior cruciate ligament reconstruction

Exclusion Criteria:

* revision surgery.
* reconstruction with a different graft from hamstring tendons.
* Associated osteotomy.
* Less than 50 kg, and allergy.
* medical contraindication for any of the components of the periarticular infiltration or postoperative analgesic medical protocol.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
Pain in the knee at 8 hours after surgery assessed by visual analog scale | registered at 8 hours
  pain registered in the knee, which was measured using a 100-mm visual analog scale from 0 (no pain) to 100 (the worst pain)
Pain in the knee at 24 hours after surgery assessed by visual analog scale | registered at 24 hours
  pain registered in the knee, which was measured using a 100-mm visual analog scale from 0 (no pain) to 100 (the worst pain)
Pain in the posterior proximal thigh at 8 hours after surgery assessed by visual analog scale | registered at 8 hours
  pain registered in the posterior proximal thigh, which was measured using a 100-mm visual analog scale from 0 (no pain) to 100 (the worst pain)
Pain in the posterior proximal thigh at 24 hours after surgery assessed by visual analog scale | registered at 24 hours
  pain registered in the posterior proximal thigh, which was measured using a 100-mm visual analog scale from 0 (no pain) to 100 (the worst pain)

SECONDARY OUTCOMES:
analgesic rescue medication | 24 hours post operative
  Number of patients who needed analgesic rescue medication in the post-anesthesia care unit and during the stay in the orthopedics ward

CONTACTS AND LOCATIONS:
Overall Officials: Joaquin De Lamo-Rovira, MD, Principal Investigator — Virgen de La Luz Hospital
Locations (1):
- Virgen de la Luz Hospital, Cuenca, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kurosaka K, Tsukada S, Nakayama H, Iseki T, Kanto R, Sugama R, Yoshiya S. Periarticular Injection Versus Femoral Nerve Block for Pain Relief After Anterior Cruciate Ligament Reconstruction: A Randomized Controlled Trial. Arthroscopy. 2018 Jan;34(1):182-188. doi: 10.1016/j.arthro.2017.08.307. Epub 2017 Dec 6. PMID 29203380
- [Background] Lefevre N, Klouche S, de Pamphilis O, Herman S, Gerometta A, Bohu Y. Peri-articular local infiltration analgesia versus femoral nerve block for postoperative pain control following anterior cruciate ligament reconstruction: Prospective, comparative, non-inferiority study. Orthop Traumatol Surg Res. 2016 Nov;102(7):873-877. doi: 10.1016/j.otsr.2016.07.011. Epub 2016 Oct 4. PMID 27720193
- [Background] Bushnell BD, Sakryd G, Noonan TJ. Hamstring donor-site block: evaluation of pain control after anterior cruciate ligament reconstruction. Arthroscopy. 2010 Jul;26(7):894-900. doi: 10.1016/j.arthro.2009.11.022. Epub 2010 May 13. PMID 20620788
- [Background] Jansson H, Narvy SJ, Mehran N. Perioperative Pain Management Strategies for Anterior Cruciate Ligament Reconstruction. JBJS Rev. 2018 Mar;6(3):e3. doi: 10.2106/JBJS.RVW.17.00059. No abstract available. PMID 29533268
- [Background] Fauno P, Lund B, Christiansen SE, Gjoderum O, Lind M. Analgesic effect of hamstring block after anterior cruciate ligament reconstruction compared with placebo: a prospective randomized trial. Arthroscopy. 2015 Jan;31(1):63-8. doi: 10.1016/j.arthro.2014.07.024. Epub 2014 Sep 17. PMID 25239172